CLINICAL TRIAL: NCT01100814
Title: Expression of S100A2 and Trefoil Factor Family Members in Epstein-Barr Virus Related Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Wei Peng Yong, National University Hospital, Singapore
Other Study IDs: GA01/08/08
Record Dates: First submitted 2009-09-15; First posted 2010-04-09 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators hypothesize that aberrant hypermethylation of tumour suppressor genes is an important mechanism for Epstein-Barr Virus (EBV) - related gastric carcinogenesis, the promoter hypermethylation status and the expression of S100A2 and TFF1 might be different between EBV-associated gastric cancer (GC) and non EBV-associated GC.

ELIGIBILITY:
Inclusion Criteria:

* Nil

Exclusion Criteria:

* Nil

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 200 gastric tumour and normal tissue samples, as well as up to 50 non-neoplastic gastric tissues samples from individuals without gastric cancer (treated for other reasons, such as gastric ulcers) will be obtained from the tissue archives of the NUH Department of Pathology. These samples were selected because relevant clinical information of these samples are available from gastric database and will allow us to perform association studies.
Sampling Method: Probability Sample
Dates: Start 2011-09; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore